CLINICAL TRIAL: NCT03154151
Title: Internet-based Psychotherapies for PTSD Symptoms in World Trade Center (WTC) Responders and Survivors
Brief Title: Online Therapy for Posttraumatic Stress Symptoms in WTC Responders and Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: National Institute for Occupational Safety and Health (NIOSH/CDC) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Adriana Feder, Associate Professor, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GCO 13-1850; U01OH010729 (NIH)
Record Dates: First submitted 2017-05-12; First posted 2017-05-16 (Actual); Last update posted 2022-01-25 (Actual); Status verified 2022-01

CONDITIONS: Post-Traumatic Stress Disorder
Keywords: PTSD; Post-Traumatic Stress Disorder; Post-Traumatic Stress Disorder symptoms; World Trade Center; 9/11; first responder; rescue/recovery/clean-up worker; trauma; 9/11 survivor
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Online Cognitive-Behavioral Therapy (Experimental): Through guided writing, Internet-based cognitive therapy aims to help WTC responders and survivors process any traumatic experiences they lived through during their WTC recovery work and exposure.
  Interventions: Behavioral: Online Cognitive-Behavioral Therapy
- Online Supportive Therapy (Active Comparator): Through guided writing, Internet-based supportive therapy aims to help WTC responders and survivors work through any life problems they might currently be experiencing.
  Interventions: Behavioral: Online Supportive Therapy

INTERVENTIONS:
Behavioral: Online Cognitive-Behavioral Therapy — Each participant will complete writing assignments focusing on how their experiences during the 9/11 attacks or the WTC recovery effort continue to affect their life, and the therapist will provide written responses and guidance within two work days, through the secure Web platform. Participants will be asked to complete one to two 45-minute writing assignments per week, over a six-week period (11 in total). Participants are asked not to begin new psychotherapy or medication with an outside therapist or doctor during the study.
  Other Names: Online Therapist-assisted Cognitive-Behavioral Therapy; Integrative Testimonial Therapy
  Arms: Online Cognitive-Behavioral Therapy
Behavioral: Online Supportive Therapy — Each participant will complete writing assignments focusing on problems and stressors that are currently affecting their life, and the therapist will provide written responses and guidance within two work days, through the secure Web platform. Participants will be asked to complete one to two 45-minute writing assignments per week, over a six-week period (11 in total). Participants are asked not to begin new psychotherapy or medication with an outside therapist or doctor during the study.
  Other Names: Online Therapist-assisted Supportive Therapy; Modified Present-Centered Therapy
  Arms: Online Supportive Therapy

SUMMARY:
If you worked or volunteered as a WTC rescue, recovery or clean-up worker after the 9/11 attacks, or are a survivor of the WTC 9/11 attacks, and you are still experiencing Posttraumatic Stress Disorder (PTSD) symptoms related to your WTC experience, you might be eligible to participate in this clinical trial of therapist-assisted, Internet-based (online) writing therapy for WTC responders and survivors with persistent PTSD symptoms. This study is for WTC responders and survivors who are not currently receiving psychotherapy/counseling. In this study, the researchers aim to find out if Internet-based therapy can help WTC responders and survivors who are still experiencing PTSD symptoms.

DETAILED DESCRIPTION:
Some people who live through traumatic experiences, such as the 9/11 WTC attacks or their aftermath, suffer from mental and physical problems that occur as a result of the incident and can persist over time. These problems are known as post-traumatic stress reactions or symptoms, and may include sleep disturbances, feelings of guilt and shame, persistent nightmares or upsetting memories of the incident, avoidance of reminders that might trigger upsetting memories, loss of interest in activities, concentration difficulties, and feeling distant from other people.

People who experience persistent PTSD symptoms often receive treatment in person in an outpatient clinic. However, recent findings suggest that Internet-based treatment can also yield positive treatment effects. The Internet offers people the opportunity to receive psychological support from home. For some people, it is easier to communicate without direct visual contact with another person about their experiences. Despite the distance, people can reflect on their situation or concerns with the help of a personal therapist.

As mentioned above, this study is for WTC responders who are not currently receiving psychotherapy/ counseling. After completing the online consent form and an initial online questionnaire, participants complete a telephone assessment conducted by a member of the team at Mount Sinai Medical Center. If you are eligible and agree to participate, you will be randomly assigned (as by the flip of a coin) to receive one of two therapies: Internet-based cognitive-behavioral therapy or Internet-based supportive therapy. Each participant is assigned a personal therapist from the team at Mount Sinai to work with throughout the treatment. In this study, communication between participant and therapist is conducted exclusively across the Internet, in written form, through the secure Web platform housed at Mount Sinai. The treatment involves written exchanges between participant and therapist over the course of approximately six weeks. Through guided writing, online therapy aims to help WTC responders process their traumatic experiences or better manage current life problems. In this study, the researchers aim to find out if Internet-based therapy can help WTC responders who are still experiencing PTSD symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Men and women who have worked or volunteered as rescue, recovery or clean-up workers at the WTC site following the 9/11 attacks, or who were living as a resident or working as an employee within the NYC disaster area during the 9/11 attacks, and who:
* are currently still experiencing significant posttraumatic stress symptoms related to what they witnessed or lived through during the 9/11 attacks or their WTC recovery work and:
* are not currently receiving psychotherapy or counseling
* do not have psychosis, a psychotic disorder, or bipolar disorder
* have not had recent alcohol or drug use problems
* are not experiencing suicidal thoughts,thoughts of harming others, or significant dissociative symptoms.

Exclusion Criteria:

* are currently taking antipsychotic medication, lithium or valproic acid.
* have a current uncontrolled medical illness, neurological disorder affecting the central nervous system, or history of head injury
* currently taking daily benzodiazepines or daily opioid medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2017-08-21 (Actual); Primary Completion 2021-05-20 (Actual); Study Completion 2021-08-10 (Actual)

PRIMARY OUTCOMES:
PTSD symptom change on the PTSD Checklist for DSM-5 | Pre- to Post-treatment, average 9 weeks
  WTC-related PTSD symptoms, assessed using total PTSD Checklist-5 (PCL-5) score. PCL-5 scores range from 0-80, with higher score indicating more severe PTSD symptoms.

SECONDARY OUTCOMES:
Durability of PTSD symptom change on the PCL-5 | 3 months post-treatment
  WTC-related PTSD symptoms, assessed using total PTSD Checklist-5 (PCL-5) score. PCL-5 scores range from 0-80, with higher score indicating more severe PTSD symptoms.
Change in PTSD symptom clusters on the PCL-5 | Pre- to Post-treatment, average 9 weeks
  PTSD symptom dimensions (DSM-5 criteria B, C, D, and E), assessed using PCL-5 subscale scores. (B) Intrusion symptoms subscale scores range from 0-20, (C) Avoidance subscale scores range from 0-8, (D) Negative alterations in cognitions and mood subscale scores range from 0-28, and (E) Alterations in arousal and reactivity subscale scores range from 0-24).
Durability of change in PTSD symptom clusters on the PCL-5 | 3 months post-treatment
  PTSD symptom dimensions (DSM-5 criteria B, C, D, and E), assessed using PCL-5 subscale scores. (B) Intrusion symptoms subscale scores range from 0-20, (C) Avoidance subscale scores range from 0-8, (D) Negative alterations in cognitions and mood subscale scores range from 0-28, and (E) Alterations in arousal and reactivity subscale scores range from 0-24).
Beck Depression Inventory II (BDI-II) | Pre- to Post-treatment, average 9 weeks
  Beck Depression Inventory II (BDI-II) is a 21-item scale for measuring the severity of depression, each item scored 0 (not present) to 3 (severe) with total from 0 (minimal depression) to 63 (severe depression).
Beck Depression Inventory II (BDI-II) | 3 months post-treatment
  Beck Depression Inventory II (BDI-II) is a 21-item scale for measuring the severity of depression, each item scored 0 (not present) to 3 (severe) with total from 0 (minimal depression) to 63 (severe depression).
GAD-7 | Pre- to Post-treatment, average 9 weeks
  Generalized Anxiety Disorder 7-item (GAD-7) scale is a 7 item scale for measuring the severity of anxiety, each item scored 0 (Not at all) to 3 (Nearly every day), with total from 0 (minimal anxiety) to 21 (severe anxiety).
GAD-7 | 3 months post-treatment
  Generalized Anxiety Disorder 7-item (GAD-7) scale is a 7 item scale for measuring the severity of anxiety, each item scored 0 (Not at all) to 3 (Nearly every day), with total from 0 (minimal anxiety) to 21 (severe anxiety).
Posttraumatic Growth Inventory - 10 Item Short Form (PTGI-SF) | Pre- to Post-treatment, average 9 weeks
  Psychological growth following a traumatic experience is assessed with the PTGI-SF. PTGI-SF is a 10-item scale for assessing positive outcomes reported by persons who have experienced traumatic events. Each item is scored 0 (did not experience) to 5 (experienced change to a great degree) with total from 0 (minimal change) to 50 (much change towards positive outcomes)
Posttraumatic Growth Inventory - 10 Item Short Form (PTGI-SF) | 3 months post-treatment
  Psychological growth following a traumatic experience is assessed with the PTGI-SF. PTGI-SF is a 10-item scale for assessing positive outcomes reported by persons who have experienced traumatic events. Each item is scored 0 (did not experience) to 5 (experienced change to a great degree) with total from 0 (minimal change) to 50 (much change towards positive outcomes)
Medical Outcomes Study Short Form 8 Health Survey | Pre- to Post-treatment, average 9 weeks
  Mental and physical functioning is assessed by the Medical Outcomes Study Short Form 8 (SF-8) Health Survey. The questions in the SF-8 target eight dimensions of health and are weighted and summed to provide two composite measures, the Physical Composite Scale and Mental Composite Scale (PCS and MCS). The PCS and MCS are scored to range from 0 to 100, with 0 indicating the lowest level of health and 100 indicating the highest level of health.
Medical Outcomes Study Short Form 8 Health Survey | 3 months post-treatment
  Mental and physical functioning is assessed by the Medical Outcomes Study Short Form 8 (SF-8) Health Survey. The questions in the SF-8 target eight dimensions of health and are weighted and summed to provide two composite measures, the Physical Composite Scale and Mental Composite Scale (PCS and MCS). The PCS and MCS are scored to range from 0 to 100, with 0 indicating the lowest level of health and 100 indicating the highest level of health.

CONTACTS AND LOCATIONS:
Overall Officials: Adriana Feder, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai; Robert H Pietrzak, PhD, MPH, Principal Investigator — Yale University
Locations (4):
- United States (4):
  - Yale University, New Haven, Connecticut
  - Boston University, Boston, Massachusetts
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - James J. Peters VA Medical Center, The Bronx, New York

IPD SHARING:
Plan to Share IPD: No